CLINICAL TRIAL: NCT05669768
Title: Study on the Efficacy and Toxicity of Pamiparib Combined With Tamoxifen in the Treatment of Epithelial Ovarian Cancer Patients With Biochemical Recurrence During First-line PARPi Maintenance Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jundong Li, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PATAOC
Record Dates: First submitted 2022-12-09; First posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pamiparib; Tamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pamiparib+tamoxifen (Experimental)
  Interventions: Drug: Pamiparib/Tamoxifen

INTERVENTIONS:
Drug: Pamiparib/Tamoxifen — Pamiparib 40mg PO BID, Tamoxifen 20mg PO BID

SUMMARY:
The goal of this phase II single arm prospective clinical study is to evaluate the efficacy and toxicity of pamiparib + tamoxifen regimen in epithelial ovarian cancer patients with biochemical recurrence during first-line PARPi maintenance therapy. The main questions it aims to answer are:

* Effect of the regimen on the reduction of CA125
* The delayed effect of treatment regimens on the patient's radiographic progression

DETAILED DESCRIPTION:
A high proportion of ovarian cancer patients tend to have elevated CA-125 2-6 months before imaging recurrence. The time between biochemical recurrence (i.e., only elevated CA125 without imaging to assess lesions or clinical symptoms) to imaging recurrence can be considered a "window period", and if imaging progression can be delayed after biochemical recurrence, the chemotherapy interval can be extended, converting platinum-resistant relapsed patients to platinum-sensitive patients, and ultimately improving patient outcomes.

The timing of treatment for these patients has been controversial, and international guidelines recommend some management approaches: 1) Follow-up observation; 2) Use of tamoxifen or other hormonal drugs; 3) Immediately administer chemotherapy according to the recurrent tumor; 4) Participate in clinical trials.

Pamiparib is a new PARPi that has shown good efficacy and safety in the posterior-line treatment of ovarian cancer patients, this study used tamoxifen combined with pamiparib to explore the efficacy and toxic side effects of this regimen in epithelial ovarian cancer patients with biochemical recurrence during first-line PARPi maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signing of the consent form;
2. Age ≥ 18 years;
3. Histologically confirmed malignant epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer, including high-grade serous cancer, low-grade serous cancer, endometrioid cancer, and clear cell cancer;
4. Patients with ovarian cancer reaching NED (no evidence of disease) or CR/PR in the last platinum containing chemotherapy after full staging or tumor cell reduction surgery (CA125 is required to be reduced to the normal range);
5. Has received first-line maintenance treatment of PARP inhibitor in the past, and the time from first-line maintenance treatment of PARP inhibitor to biochemical recurrence is required to be ≥ 12 months;
6. The type of PARP inhibitor used in the past is not limited, and it is allowed to change the type of PARP inhibitor due to non disease progression;
7. CA-125 increased more than twice the upper limit of normal value again, but imaging examination showed no evidence of tumor recurrence;
8. The expected life span is more than 3 months;
9. The ECOG score of the Eastern Tumor Cooperation Group was 0-1;
10. The main organs function well, which is defined as:

    * Absolute neutrophil count (ANC) ≥ 1.5 × 10L
    * Platelet count (PLT) ≥ 75 × 10L
    * Hemoglobin ≥ 9gdL
    * Serum creatinine Cr<1.5 × Upper limit of normal value (ULN)
    * Total serum bilirubin ≤ 1.5 × Upper limit of normal range (ULN)
    * Both glutamic oxaloacetic transaminase and glutamic pyruvic transaminase ≤ 3XULN
    * Coagulation function: international standardized ratio (NR) ≤ 1.5; When activated partial prothrombin (APTT) ≤ 1.5XULN, prophylactic use of low-dose aspirin and low-molecular-weight heparin is allowed;
11. If the patient has been tested for g/tBRCA1/2 gene in the past, the corresponding test report shall be provided; If the g/tBRCA1/2 gene test has not been performed in the past, it is necessary to provide archived tumor tissue samples (formalin fixed, paraffin embedded tumor tissue blocks) or fresh tumor tissue samples for making at least 5 tissue sections for BRCAm test (optional)

Exclusion Criteria:

1. Patients with other malignant tumors (except for patients with carcinoma in situ who have been fully treated and have no disease evidence, except for patients with thyroid cancer who have completed radical treatment, and patients with other malignant tumors who have completed radical treatment and have been screened for more than 5 years from the last tumor related treatment);
2. Imaging evaluation showed clear evidence of tumor recurrence or progression;
3. Pregnancy and perinatal patients;
4. Active pneumonia not cured;
5. History of important organ transplantation;
6. History of serious mental illness and brain dysfunction;
7. Drug abuse or drug abuse history;
8. Any active autoimmune disease or patient with a history of autoimmune disease (including but not limited to autoimmune hepatitis, interstitial pneumonia, hepatitis, enteritis, nephritis, hypophysitis, vasculitis, uveitis) or patients who need systemic hormone therapy and/or immunosuppression therapy (such as asthma requiring bronchodilators); Except for the following: vitiligo, alopecia, Graves syndrome, psoriasis or eczema that do not need systematic treatment in the past 2 years, stable immune thyroiditis that has been controlled after treatment, type I diabetes that only needs stable insulin, and childhood asthma has been completely alleviated;
9. The immunosuppressant or systemic hormone therapy is being used to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other equivalent hormone preparations), and it is still used 2 weeks before enrollment. Local and systemic use of prednisone or other equivalent hormone preparations not exceeding 10mg/day is allowed;
10. Patients with active bleeding (bleeding caused by tumor needs to be evaluated by the researcher), bleeding tendency or risk of massive bleeding (such as tumor involving large vessels, important bronchi, obvious bleeding beyond control after hemostasis treatment, and uncured bronchiectasis), or patients who need to be treated with coumarin anticoagulants at the same time;
11. Thrombosis or embolism events occurred in the past 6 months, such as cerebrovascular accident (including transient ischemic attack);
12. Serious cardiovascular disease or medical history includes but is not limited to the following:

    * NYHA Grade 3 and 4 congestive heart failure within 6 months before enrollment
    * Unstable angina or newly diagnosed angina or myocardial infarction within 12 months before screening
    * Arrhythmias requiring treatment intervention (Patients with administration of β- receptor blockers or digoxin can be enrolled)
    * Family history of prolonged QT interval syndrome or corrected QT interval (QTc)>450ms; If the patient has an extended QTc interval, but the reason assessed by the investigator is that the pacemaker (and there is no other cardiac abnormality) is still included in the group
    * CTCAE ≥ Grade 2 valvular heart disease
    * Hypertension with poor control (systolic blood pressure>150 mmHg or diastolic blood pressure>100 mmHg;
13. Patients with moderate or above pulmonary dysfunction and unable to relieve them have interstitial lung disease or active pulmonary tuberculosis;
14. Patients with active ulcer, intestinal perforation, unresponsive intestinal obstruction, and patients with a history of gastrointestinal perforation within 28 days before inclusion in the study;
15. Active inflammatory bowel disease, uncontrollable nausea and vomiting, inability to swallow the study drug, and any gastrointestinal disease that may interfere with drug absorption and metabolism;
16. Active infections such as human immunodeficiency virus, syphilis, and untreated active hepatitis (HBV DNA copy number is greater than 1000 IU/ml, and HCV RNA is positive);
17. Serious infection occurred 4 weeks before the first administration;
18. Other serious or uncontrollable diseases, including but not limited to:

    * Uncontrolled grand mal, unstable spinal cord compression, superior vena cava syndrome or other mental disorders that affect the patient's informed consent;
    * Immune deficiency (excluding splenectomy), or other diseases that the researcher thinks may expose the patient to high risk toxicity;
    * Those who have a history of abuse of psychotropic substances and are unable to quit or have mental disorders;
19. Inoculate live vaccine or attenuated live vaccine 30 days before the first administration;
20. Known allergy to active or inactive ingredients of the study drug or drugs with similar chemical structure; Patients who are pregnant or nursing, or who are expected to become pregnant during the study treatment;
21. Other laboratory inspection abnormalities:

    * Uncorrectable hyponatremia (sodium<130 mmol/L; serum potassium<3.5 mmol/L)
    * Any past or current disease, treatment or laboratory abnormality that may interfere with the results of the study and affect the patient's participation in the study, or the investigator believes that the patient is not suitable to participate in the study;
22. Any situation that the researcher thinks is not suitable for participating in the research, including poor understanding and low cooperation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Response rate by CA-125 | Up to approximately 24 months
  Best overall response in patients without initial measurable disease and who are evaluable by CA 125 is according to the Gynecological Cancer Intergroup (GCIG)

SECONDARY OUTCOMES:
PFS (progression-free survival) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  PFS of parmiparib in combination with tamoxifen in epithelial ovarian cancer patients with biochemical recurrence during first-line PARPi maintenance therapy was assessed by investigators according to RECIST v1.1
TFST (Time to first subsequent therapy) | TFST was defined as the time from the onset of patient enrollment to the time of first subsequent treatment or death, whichever occurs first, up to 24 months.
  TFST of parmiparib in combination with tamoxifen in epithelial ovarian cancer patients with biochemical recurrence during first-line PARPi maintenance therapy was assessed by investigators according to the time when the patients started subsequent treatment
The percentage of subjects discontinued study treatment due to adverse events assessed according to NCI-CTCAE v5.0. | Up to approximately 24 months
  Safety and tolerability
EORTC-QLQ-C30（EORTC Core Quality of Life questionnaire） | Up to approximately 24 months
  The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire assesses important functioning domains (e.g. physical, emotional, role) and common cancer symptoms (e.g. fatigue, pain, nausea/vomiting, appetite loss).
  The EORTC QLQ-C30 was scored according to the scoring manual. This produced scores on 15 subscales (range for each, 0-100), with higher scores indicating better outcomes on global quality of life/health and functioning subscales and worse outcomes on symptom scales and for financial problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Centre, Guangzhou, Guangdong, China